CLINICAL TRIAL: NCT00490672
Title: Community Based Multiple Risk Factors Intervention Strategy to Prevent Cardiovascular and Chronic Kidney Diseases [CORFIS]
Brief Title: Community Based Multiple Risk Factors Intervention Strategy
Acronym: CORFIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ministry of Health, Malaysia (Other Government)
Responsible Party: Dr. Lim Teck Onn, Clinical Research Centre, Hospital Kuala Lumpur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT07-02; NMRR ID Number: 447
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2010-04

CONDITIONS: Hypertension; Diabetes Mellitus; Hyperlipidemia
Keywords: Hypertension; Diabetes Mellitus; Hyperlipidaemia; Primary Care; Community Care; Multiple Risk Factors Interventional Strategies
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Hyperlipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Arm (Other): Conventional Patient Management on Hypertension, Diabetes Mellitus and Hyperlipidaemia by Malaysian GP
  Interventions: Behavioral: No Active Intervention.
- CORFIS Arm (Active Comparator): Community based Multiple Risk Factor Intervention Strategies
  Interventions: Behavioral: Community Based Multiple Risk Factor Intervention Strategies

INTERVENTIONS:
Behavioral: No Active Intervention. — Conventional Chronic Disease Management in Malaysia Primary Care
  Other Names: Control
  Arms: Control Arm
Behavioral: Community Based Multiple Risk Factor Intervention Strategies — Multi-faceted Intervention in Chronic Diseases Management i.e. Hypertension, Diabetes Mellitus, Hyperlipidaemia involving Primary Health Care Physicians, Nurse Educators, Dieticians and Pharmacists.
  Other Names: CORFIS
  Arms: CORFIS Arm

SUMMARY:
Randomized controlled trial of CORFIS Programme.

The study objectives are as follows:

1. To determine the efficacy of a community based multiple risk factors interventional strategy (CORFIS) for a treatment period of 6 months in patients on treatment for HT, DM or HL.
2. The intervention shall consist of a purpose design and systematically organized disease management program that employ multi-faceted interventions incorporating various specific measures to maximize both clinician (as investigator) adherence with treatment guideline and patient adherence with treatment.

DETAILED DESCRIPTION:
It should be obvious to all that we urgently need to improve the management of the various risk factors for cardiovascular (CVD) and chronic kidney diseases (CKD); the 3 most important of which are Hypertension (HT), Diabetes mellitus (DM), Hyperlipidaemias (HL). It is not just that these are highly prevalent in our community, they are also poorly managed and controlled, with resulting highly costly and adverse health impact on our population. It should also be equally obvious that we need a better approach to manage these risk factors in our community. There have been considerable advances in our understanding of these risk factors and in our knowledge of the variety of approaches to achieving control of these risk factors including the role of self-monitoring and self-management education, medical nutrition therapy, physical activity, psychological counseling, and various drug therapy options.

This study is a multi-center, open label, parallel group randomized trial designed to demonstrate the effectiveness of a community based multiple risk factors interventional strategy (CORFIS).

750 patients on treatment for HT, DM or HL from 75 general practices (GPs) who meet inclusion/exclusion criteria will be enrolled into the trial. Among the 75 selected GPs, 50 of them will be randomly allocated to CORFIS and 25 to routine care.

After initial screening, patients will attend clinic for baseline examination. Study prescribed visits for efficacy and safety assessments will occur monthly for 6 months. Hence there will be a total of 7 visits.

ELIGIBILITY:
Inclusion criteria:

1. Patients diagnosed by participating GP to have Hypertension and/or Diabetes mellitus and/or Hyperlipidaemias, and currently on drug treatment for one or more of these conditions
2. Patients age 18 years and above.
3. Written informed consent obtained from patients.

Exclusion criteria:

1. Pregnant or nursing women.
2. History of unstable angina, acute myocardial infarction or coronary revascularisation procedure in the preceding 6 months.
3. Clinically significant valvular heart disease.
4. Overt heart failure or history of heart failure in the preceding 6 months
5. Stroke in the preceding 6 months.
6. Serum creatinine more than 150umol/l in the preceding 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients able to reach treatment goals. | 6 months follow up

SECONDARY OUTCOMES:
The safety of the drug product used in the study will be assessed using the procedure for adverse drug reactions reporting for marketed medicinal products regulated by the Malaysian regulatory authority. | 6 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Teck Onn Lim, FRCP, Principal Investigator — Ministry of Health, Malaysia; Zaki M Mohd Zaher, FRCP, Study Chair — International Medical University Malaysia
Locations (78):
- Malaysia (78):
  - Klinik Dr Khalil, Kuala Lumpur, Federal Territoy
  - Horeb Sdn Bhd, Kuala Lumpur, Kuala Lumpur
  - Klinik Tan & Mano Sdn Bhd, Kuala Lumpur, Kuala Lumpur
  - Klinik Kaulsay, Kuala Lumpur, Kuala Lumpur
  - Klinik Unimed Plaza Damansara, Kuala Lumpur, Kuala Lumpur
  - Poliklinik Kumpulan City (Plaza Damansara), Kuala Lumpur, Kuala Lumpur
  - Klinik Shafi, Kuala Lumpur, Kuala Lumpur
  - Poliklinik Kepong Baru, Kuala Lumpur, Kuala Lumpur
  - Klinik Chew, Kuala Lumpur, Kuala Lumpur
  - Klinik Reddy Setapak, Kuala Lumpur, Kuala Lumpur
  - Klinik Medik (Dr Amir & Rakan-Rakan), Kuala Lumpur, Kuala Lumpur
  - Klinik Keluarga, Kuala Lumpur, Kuala Lumpur
  - Klinik Vicky, Kuala Lumpur, Kuala Lumpur
  - Klinik Care Poliklinik & Surgeri, Kuala Lumpur, Kuala Lumpur
  - Klinik Tenaga Baru, Kuala Lumpur, Kuala Lumpur
  - Kumpulan Medi-Systems Sdn Bhd, Kuala Lumpur, Kuala Lumpur
  - Poliklinik Salak Selatan, Kuala Lumpur, Kuala Lumpur
  - Klinik Sharon, Kuala Lumpur, Kuala Lumpur
  - Klinik Medi Pesona, Kuala Lumpur, Kuala Lumpur
  - Klinik Sharani, Kuala Lumpur, Kuala Lumpur
  - Klinik Prime Care, Kuala Lumpur, Kuala Lumpur
  - PoliKlinik Bangsar, Kuala Lumpur, Kuala Lumpur
  - Poliklinik Medics, Kuala Lumpur, Kuala Lumpur
  - Klinik Famili TTDI, Kuala Lumpur, Kuala Lumpur
  - Klinik Ehsan, Mentakab, Pahang
  - Klinik Dan Surgeri Putra, Ampang, Selangor
  - Klinik Idzham Sdn Bhd, Ampang, Selangor
  - Klinik Mediviron, Ampang, Selangor
  - Klinik Putera (Poliklinik Bistari), Ampang, Selangor
  - Klinik Tan & Mano, Ampang, Selangor
  - Poliklinik Gomez 24 Jam, Ampang, Selangor
  - Poliklinik Penawar, Ampang, Selangor
  - Klinik Hayati (Poliklinik & Surgeri), Batu Caves, Selangor
  - Klinik Nathan Dan Rakan-Rakan, Batu Caves, Selangor
  - Poliklinik Idaman, Batu Caves, Selangor
  - Poliklinik Kumpulan City, Batu Caves, Selangor
  - MAS Medical Centre, Kampung Baru Subang, Selangor
  - Klinik Keluarga Azian & Elina, Klang, Selangor
  - Klinik Keluarga Siva Lim, Klang, Selangor
  - Lok Dispensary, Klang, Selangor
  - Klinik Bandaran, Klang, Selangor
  - Klinik Kelang, Klang, Selangor
  - Klinik Lim, Klang, Selangor
  - Klinik Yuen, Klang, Selangor
  - Klinik Stella Maris Sdn Bhd, Klang, Selangor
  - Klinik Utama, Klang, Selangor
  - Klinik Wan Elina, Klang, Selangor
  - Poliklinik Hari, Klang, Selangor
  - Klinik Ng & Lim, Klang, Selangor
  - Klinik Khaty Am, Petaling Jaya, Selangor
  - Poliklinik Shaik (Sunway) Sdn Bhd, Petaling Jaya, Selangor
  - Klinik Primecare, Petaling Jaya, Selangor
  - Klinik Petaling Jaya, Petaling Jaya, Selangor
  - Klinik Alam Medic, Petaling Jaya, Selangor
  - Klinik Rakan Medik, Petaling Jaya, Selangor
  - Poliklinik Rakyat, Petaling Jaya, Selangor
  - Klinik Kelana Puteri, Petaling Jaya, Selangor
  - Klinik Ready Care, Petaling Jaya, Selangor
  - Poliklinik Hidayah, Petaling Jaya, Selangor
  - Klinik Dr Shamsuddin, Petaling Jaya, Selangor
  - Klinik Hafiz, Puchong, Selangor
  - Klinik Leong, Puchong, Selangor
  - Klinik Raya, Puchong, Selangor
  - Klinik Reddy, Puchong, Selangor
  - Klinik Ng Singh & Rakan-Rakan, Rawang, Selangor
  - Klinik Sarrimadh, Seri Kembangan, Selangor
  - Klinik Bandaran Sdn Bhd, Shah Alam, Selangor
  - Klinik Kelang, Shah Alam, Selangor
  - Poliklinik Sri Muda, Shah Alam, Selangor
  - Klinik Dan Surgeri Alpha Medic, Shah Alam, Selangor
  - Klinik Medic Bestari, Subang Jaya, Selangor
  - Klinik Medifom, Subang Jaya, Selangor
  - Victor Medical Practice, Subang Jaya, Selangor
  - Klinik Medijaya, Subang Jaya, Selangor
  - Klinik Dr Nur Ainita, Subang Jaya, Selangor
  - Klinik Taipan, Subang Jaya, Selangor
  - Poliklinik Roshan, Subang Jaya, Selangor
  - Klinik Kok dan Wendy, Subang Jaya, Selangor

REFERENCES:
- [Derived] Chua SS, Kok LC, Yusof FA, Tang GH, Lee SW, Efendie B, Paraidathathu T. Pharmaceutical care issues identified by pharmacists in patients with diabetes, hypertension or hyperlipidaemia in primary care settings. BMC Health Serv Res. 2012 Nov 12;12:388. doi: 10.1186/1472-6963-12-388. PMID 23145922